CLINICAL TRIAL: NCT01916681
Title: Foley OR MisO for the Management of Induction (FOR MOMI) Trial
Brief Title: Foley OR MisO for the Management of Induction
Acronym: FORMOMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 817897
Record Dates: First submitted 2013-07-30; First posted 2013-08-06 (Estimated); Results first posted 2016-12-21 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-04

CONDITIONS: Delivery; Prolonged
Keywords: Induction; Labor; Cervical foley; Misoprostol; Pitocin; Oxytocin; Cytotec; Delivery; IOL
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cervical foley & Misoprostol (Experimental): Patients randomized to this arm will receive a cervical foley and misoprostol to induce their labor.
  Interventions: Device: Cervical Foley & Misoprostol
- Misoprostol only (Experimental): Patients randomized to this arm will receive misoprostol only to induce their labor.
  Interventions: Drug: Misoprostol Alone
- Cervical foley alone (Experimental): Patients randomized to this arm will receive a cervical foley to induce their labor.
  Interventions: Device: Cervical Foley Alone
- Cervical foley & Pitocin (Experimental): Patients randomized to this arm will receive a cervical foley and pitocin to induce their labor.
  Interventions: Device: Cervical Foley & Pitocin

INTERVENTIONS:
Device: Cervical Foley & Misoprostol — A cervical foley combined with misoprostol will be used to induce the patient.
  Other Names: Misoprostol is also known as Cytotec
  Arms: Cervical foley & Misoprostol
Drug: Misoprostol Alone — Misoprostol will be used alone to induce the patient
  Other Names: Misoprostol is also known as Cytotec
  Arms: Misoprostol only
Device: Cervical Foley Alone — A cervical foley alone will be used to induce the patient
  Arms: Cervical foley alone
Device: Cervical Foley & Pitocin — A cervical foley combined with pitocin will be used to induce the patient
  Other Names: Pitocin is also known as Oxytocin
  Arms: Cervical foley & Pitocin

SUMMARY:
The percentage of women undergoing an induction of labor (IOL) is estimated to be 20% and continues to rise. Simultaneously, the cesarean delivery (CD) rate has continued to increase (2). Induction is a known risk factor for CD. Despite numerous studies evaluating time periods to define a failed IOL, there are no guidelines or accepted definitions of when to call an IOL failed given the incremental gain in vaginal delivery when IOL is prolonged. While decreasing the CD rate is an important primary focus in obstetrics, attention must also be paid to the overall length of labor given that prolonged labor is associated with adverse maternal and neonatal outcomes. Furthermore, a prolonged labor is associated with an increase in direct hospital costs and healthcare utilization. The use of cervical ripening agents, such as vaginal prostaglandin and mechanical dilators, has been demonstrated to reduce labor time and CD rate. In addition to specific individual agents, certain dosing and regimens for IOL and active labor have been compared to evaluate whether a particular dose or regimen can decrease the length of labor and decrease the CD rate. Most of these regimens; however, focus on individual induction agents and few have compared the efficacy of using more than one agent simultaneously. Given the associated risks of prolonged labor and limited data evaluating the use of combined cervical ripening agents, our objective is to evaluate the difference in time to delivery among women who undergo an IOL with four different methods.

DETAILED DESCRIPTION:
Prolonged labor increases the risk of maternal and neonatal morbidity as well as increases healthcare costs. There is limited data evaluating the use of two simultaneous induction agents to decrease the time to delivery.

1. Maternal and neonatal morbidity with prolonged labor The adverse maternal and neonatal morbidity association with prolonged labor has been demonstrated in numerous studies. An increase in maternal risk of post partum hemorrhage and endometritis has been associated with prolonged labor. Cheng et al demonstrated that the risk of post partum hemorrhage and endometritis significantly increased with increasing length of labor. Maghoma et al evaluated the latent phase of labor and found a similar increased risk in endometritis but also noted a significant risk in maternal sepsis with a prolonged latent phase of labor.

   Neonatal outcomes are similarly improved with a shorter duration of labor. In addition to the risk of chorioamnionitis and decreased 5 minute Apgar score, there is also a significantly increased risk of neonatal intensive care unit admission as well as neonatal sepsis with prolonged labor.
2. Increased healthcare utilization with prolonged labor Both direct and indirect medical costs have been evaluated in the obstetrics literature. A prolonged labor has been associated with an increase in direct and indirect medical costs as well as an increase in healthcare utilization. Mackenzie et al evaluated the cost of different induction regimens and found a decreased cost for women that remained on the antenatal unit for a shorter period of time.
3. Use of simultaneous induction agents Pettker et al evaluated the use of a transcervical foley with and without oxytocin and found no difference in mode of delivery or delivery within 24 hours. They found that labor was 2.5 hours shorter with the addition of oxytocin although the study was not powered to see a statistical difference. Other studies have looked at the concurrent use of prostaglandin with cervical foley. Barrilleaux et al evaluated the use of oral misoprostol with cervical foley compared to cervical foley alone and found no difference in time to delivery; however, the use of oral misprostol has well known side effects, including a high rate of tachysystole which was found in this study. Hill et al reported a decreased time to second stage and time to delivery with the use of cervical foley and oral misoprostol compared to vaginal misoprostol alone; however this was a small study that used with a higher, more favorable starting Bishop score in the combined foley+misoprostol group, biasing them away from the null. Standardized time cut offs during IOL were not used in this study. Recently, Carbone et al performed a randomized trial comparing foley bulb and misprostol to misoprostol alone and found a decreased time to delivery among those in the combined group. This study was a small trial with 60 patients in each arm and did not compare the combined agents to cervical foley alone.
4. Standardization of IOL The optimal length for an IOL is not well established and data on definitions of a failed IOL and prolonged latent phase are lacking. Multiple studies have shown that within 6 hours of oxytocin administration, 60-70% of patients are in active labor. Although data suggest that the longer latent labor is allowed to proceed, the more women that will deliver vaginally, there is also evidence of an increased risk of morbidity, without a large incremental gain. Certain dosing and regimens of individual agents have been evaluated to try and decrease labor; however, studies have not evaluated the use of time cut offs during an IOL to help reduce variation in practice and standardize the IOL process.

ELIGIBILITY:
Inclusion Criteria:

* All women 18 years of age or greater
* singleton gestation
* vertex presentation
* 37 weeks gestational age or greater
* undergoing an IOL
* bishop score less than or equal to 6
* cervical dilation less than or equal to 2cm

Exclusion Criteria:

* All women less than 18 years of age
* Contraindication for vaginal delivery
* Prior cesarean delivery
* Multiple gestation
* Intrauterine fetal demise
* Fetal anomaly
* HIV
* Unable to consent/ non-English speaking
* Non-reassuring fetal heart rate
* Patients with hemolysis elevated liver enzymes and low platelets
* Eclampsia
* Intrauterine growth restriction (IUGR) 5th percentile with abnormal dopplers
* IUGR less than 10th percentile with reversed end diastolic flow
* Recurrent late decelerations w
* Continuous contractions more than 3 times in 10 minutes at onset of IOL (given that this is a contraindication to misoprostol use at our institution)
* Bishop score is greater than 6
* Cervical dilation greater than or equal to 2cm
* Confirmed ruptured membranes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 2013-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa D Levine, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- [Derived] Levine LD, Downes KL, Elovitz MA, Parry S, Sammel MD, Srinivas SK. Mechanical and Pharmacologic Methods of Labor Induction: A Randomized Controlled Trial. Obstet Gynecol. 2016 Dec;128(6):1357-1364. doi: 10.1097/AOG.0000000000001778. PMID 27824758

RESULTS

PARTICIPANT FLOW:
Groups:
- Misoprostol Only: Patients randomized to this arm will receive misoprostol to induce their labor.
  Misoprostol Alone: Misoprostol will be used alone to induce the patient
- Cervical Foley & Pitocin: Patients randomized to this arm will receive a cervical foley and pitocin to induce their labor.
  Cervical Foley & Oxytocin: A cervical foley combined with oxytocin will be used to induce the patient
Period: Overall Study
Arm/Group | Cervical Foley & Misoprostol | Misoprostol Only | Cervical Foley Alone | Cervical Foley & Pitocin
Started | 123 | 120 | 123 | 125
Completed | 123 | 120 | 123 | 125
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervical Foley & Misoprostol | Misoprostol Only | Cervical Foley Alone | Cervical Foley & Pitocin | Total
Number analyzed (Participants) | 123 | 120 | 123 | 125 | 491
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 123 | 120 | 123 | 125 | 491
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 28 [22.4 to 33.1] | 26.7 [21.8 to 31.0] | 27.3 [22.3 to 32.9] | 26.5 [22.4 to 31.7] | 27 [22 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 120 | 123 | 125 | 491
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 123 | 120 | 123 | 125 | 491

OUTCOME MEASURES:

1. Primary Outcome: Time to Delivery
Description: Amount of hours that pass between the start of the induction to delivery.
Time Frame: Hours between start of induction to delivery
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Cervical Foley & Misoprostol | Misoprostol Only | Cervical Foley Alone | Cervical Foley & Pitocin
Number analyzed (Participants) | 123 | 120 | 123 | 125
Hours | 13.1 [9.1 to 18.3] | 17.6 [11.9 to 26.7] | 17.7 [12.6 to 24.9] | 14.5 [9.3 to 20.0]

2. Primary Outcome: Length of Stay
Description: Total maternal length of stay as defined as days from the day the induction began to the day of discharge
Time Frame: Days between admit to hospital and discharge
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Cervical Foley & Misoprostol | Misoprostol Only | Cervical Foley Alone | Cervical Foley & Pitocin
Number analyzed (Participants) | 123 | 120 | 123 | 125
Days | 3 [3 to 4] | 3 [3 to 4] | 3 [3 to 4] | 3 [3 to 4]

3. Primary Outcome: Severe RDS
Time Frame: enrollment through neonatal discharge
Measure: Number; unit: participants
Arm/Group | Cervical Foley & Misoprostol | Misoprostol Only | Cervical Foley Alone | Cervical Foley & Pitocin
Number analyzed (Participants) | 123 | 120 | 123 | 125
participants | 0 | 1 | 2 | 0

4. Secondary Outcome: Mode of Delivery
Description: Cesarean Delivery
Time Frame: Start of induction to delivery
Measure: Number; unit: participants
Arm/Group | Cervical Foley & Misoprostol | Misoprostol Only | Cervical Foley Alone | Cervical Foley & Pitocin
Number analyzed (Participants) | 123 | 120 | 123 | 125
participants | 34 | 29 | 35 | 38

5. Secondary Outcome: Time to Active Labor
Time Frame: Start of induction to active labor
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Cervical Foley & Misoprostol | Misoprostol Only | Cervical Foley Alone | Cervical Foley & Pitocin
Number analyzed (Participants) | 123 | 120 | 123 | 125
Hours | 7.4 [4.4 to 10.7] | 13.3 [9.1 to 22.4] | 11.0 [7.9 to 14.9] | 8.1 [5.3 to 11.2]

6. Secondary Outcome: Regional Anesthesia
Time Frame: During delivery
Measure: Number; unit: participants
Arm/Group | Cervical Foley & Misoprostol | Misoprostol Only | Cervical Foley Alone | Cervical Foley & Pitocin
Number analyzed (Participants) | 123 | 120 | 123 | 125
participants | 114 | 111 | 114 | 121

7. Secondary Outcome: Chorioamnionitis
Time Frame: Enrollment through deischarge
Measure: Number; unit: participants
Arm/Group | Cervical Foley & Misoprostol | Misoprostol Only | Cervical Foley Alone | Cervical Foley & Pitocin
Number analyzed (Participants) | 123 | 120 | 123 | 125
participants | 15 | 9 | 17 | 20

8. Secondary Outcome: Maternal Morbidity
Time Frame: Enrollment through discharge
Measure: Number; unit: participants
Arm/Group | Cervical Foley & Misoprostol | Misoprostol Only | Cervical Foley Alone | Cervical Foley & Pitocin
Number analyzed (Participants) | 123 | 120 | 123 | 125
participants | 5 | 8 | 13 | 10

ADVERSE EVENTS:
Time Frame: Up to 6 weeks postpartum.
Arm/Group | Cervical Foley & Misoprostol | Misoprostol Only | Cervical Foley Alone | Cervical Foley & Pitocin
Serious Adverse Events (participants affected / at risk) | 0/123 | 0/120 | 0/123 | 0/125
Other Adverse Events (participants affected / at risk) | 30/123 | 33/120 | 46/123 | 46/125
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervical Foley & Misoprostol (N=123) | Misoprostol Only (N=120) | Cervical Foley Alone (N=123) | Cervical Foley & Pitocin (N=125)
Chorioamnionitis (Pregnancy, puerperium and perinatal conditions) | 15 (15) | 9 (9) | 17 (17) | 20 (20) — Defined by use of antibiotics during labor not for GBS+ or other known infection.
Endometritis (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Diagnosed and treated based on maternal fever (>100.4) in the setting of either (1) fundal tenderness or (2) maternal tachycardia
Wound Infection (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 1 (1) | 3 (3) — Diagnosed on chart review by provider documenting a diagnosis of cellulitis, need for antibiotics to treat wound, wound separation, purulent discharge from wound, abscess, or need for debridement.
Venous Thromboembolism (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Maternal blood transfusion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 5 (5) | 4 (4)
Postpartum readmission (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2) | 3 (3) | 7 (7)
NICU admission (Pregnancy, puerperium and perinatal conditions) | 10 (10) | 15 (15) | 17 (17) | 11 (11)
Neonatal blood transfusion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxic-ischemic encephalopathy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraventricular hemorrhage Grade 3 or 4 (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Severe respiratory distress (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 2 (2) | 0 (0) — Intubation and mechanical ventilation for a minimum of 12 hours.
Necrotizing enterocolitis or rule out NEC (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Culture proven neonatal sepsis (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presumed Sepsis (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No